CLINICAL TRIAL: NCT00002444
Title: Phase I/II Open Label Evaluation of Nitazoxanide for the Treatment of Cryptosporidiosis in AIDS Patients
Brief Title: A Study of Nitazoxanide in the Treatment of AIDS-Related Diarrhea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unimed Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 253A; UMD-95-004
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide

SUMMARY:
To determine the pharmacokinetics profile of single doses of nitazoxanide (NTZ) in patients with AIDS-related cryptosporidial diarrhea. To determine steady state concentrations of NTZ following repeated dosing. To assess the safety and efficacy of 4 dose levels of NTZ in these patients.

Cryptosporidial enterocolitis in AIDS patients is frequently chronic and severe, contributing substantially to morbidity, mortality, and health care costs in this population. NTZ exhibits antimicrobial activity that may extend to Cryptosporidial infection.

DETAILED DESCRIPTION:
Cryptosporidial enterocolitis in AIDS patients is frequently chronic and severe, contributing substantially to morbidity, mortality, and health care costs in this population. NTZ exhibits antimicrobial activity that may extend to Cryptosporidial infection.

Patients are enrolled in groups of 7. Group A receives the lowest dose of NTZ. Groups B - D receive sequentially higher doses. Patients in Groups B - D do not begin therapy until all patients have been enrolled at the preceding dose. For determination of single-dose pharmacokinetics, patients receive a single dose of NTZ on Day 1 and blood samples are obtained over the next 24 hours. Immediately following the 24-hour blood sample collection, patients begin the treatment phase during which they take NTZ for an additional 13 days. Blood samples are obtained again on Day 14 to determine full plasma concentration-time profiles over the dosing interval. At the end of treatment, responders discontinue treatment and nonresponders continue NTZ treatment for an additional 14 days on the same dose. Patients who still fail to respond are provided with an additional month of NTZ. Patients have scheduled visits for clinical and parasitologic efficacy assessments and safety laboratory tests.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* AIDS diagnosis according to CDC criteria.
* CD4 count less than or equal to 200 cells/mm3 or CD4 count greater than or equal to 200 cells/mm3 and documented cryptosporidiosis for a minimum of 4 weeks.
* Cryptosporidial diarrhea as defined by:
* (1) presence of Cryptosporidium oocytes in a stool specimen within 14 days of enrollment; and (2) chronic diarrhea (i.e., an average of at least 4 bowel movements per day for a minimum of 2 weeks).
* Life expectancy of at least 1 month.
* Ability to tolerate food by mouth.

Prior Medication:

Required:

* Any anti-diarrheal or anti-emetic medication for which the dosage regimen has been stable for at least 1 week prior to enrollment.
* Any antiretroviral medications (e.g., zidovudine, ddI, ddC) for which the dosage regimen has been stable for at least 3 weeks prior to enrollment.

Allowed:

Medication for prophylaxis or maintenance therapy of opportunistic infection, stable for at least 2 weeks prior to enrollment.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

Grade 4 (hematologic) or Grade 3 (for all others) toxicity. (Patients with Grade 3 toxicity for hepatic parameters may be enrolled if, in the investigator's judgment, the abnormalities are due to biliary cryptosporidiosis.)

Patients with the following prior conditions are excluded:

* Presence of Salmonella, Shigella, Campylobacter, Yersinia, Giardia lamblia, Entamoeba histolytica, Microsporidia, Isospora, Cyclospora, or Clostridium difficile toxin in stool (based on assessment within 14 days prior to enrollment by stool ova and parasite examination, culture, and C. difficile assay).
* History of intestinal Mycobacterium avium intracellular infection or intestinal Kaposi's sarcoma.
* History of Cytomegalovirus colitis, unless 28 days of therapy with ganciclovir or foscarnet completed subsequent to diagnosis.

Prior Medication:

Excluded:

* Investigational drug therapy within 14 days of enrollment, unless available under an FDA-authorized expanded access program.
* Any drug or therapy with possible anticryptosporidial activity (e.g., paromomycin, spiramycin, azithromycin, clarithromycin, hyperimmune bovine colostrum) within 14 days of enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 1995-10; Study Completion 1996-02

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Soave, Principal Investigator
Locations (1):
- New York Hosp / Cornell Med Ctr, New York, New York, United States

REFERENCES:
- [Derived] Mazzoni S, Hill P, Briggs A, Barbier K, Cahill A, Macones G, Colditz G, Tuuli M, Carter E. The effect of group prenatal care for women with diabetes on social support and depressive symptoms: a pilot randomized trial. J Matern Fetal Neonatal Med. 2020 May;33(9):1505-1510. doi: 10.1080/14767058.2018.1520832. Epub 2018 Sep 25. PMID 30251569